CLINICAL TRIAL: NCT06555393
Title: A Preliminary Human Study on Bioavailability and Efficacy of Bioactive Peptide IRW in Egg White Hydrolysate
Brief Title: Understanding the Health Effect of a Bioactive Peptide From Egg: A Pilot Study
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00125956
Record Dates: First submitted 2024-08-12; First posted 2024-08-15 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: High Blood Sugar; High Blood Pressure; Overweight and Obesity
Keywords: high blood pressure; high blood sugar; overweight; obesity
MeSH Terms: conditions — Hyperglycemia; Hypertension; Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Double-blind randomized cross-over study.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Egg white powder (20g) (Placebo Comparator): 20 g of egg white powder from the market; negative control; only individuals at risk of diabetes/having type 2 diabetes.
  Interventions: Dietary Supplement: Egg White Powder
- Egg white hydrolysate Thermoase (5 g) (powder) (Experimental): 5 g; dose based on human equivalent dose calculation; only individuals at risk of diabetes/having type 2 diabetes
  Interventions: Dietary Supplement: Egg White Powder
- Egg white hydrolysate Thermoase (20 g) (powder) (Experimental): 20 g; dose based on energy percentage used in animal experiment; both healthy control group and at risk of diabetes/having type 2 diabetes
  Interventions: Dietary Supplement: Egg White Powder
- Egg white hydrolysate Thermoase + Pepsin (20 g) liberating IRW (powder) (Active Comparator): 20 g; positive control, only individuals at risk of diabetes/having type 2 diabetes
  Interventions: Dietary Supplement: Egg White Powder

INTERVENTIONS:
Dietary Supplement: Egg White Powder — Participants will consume a standardized breakfast (2 slices of 70 g whole wheat bread, 10 g of butter and 30 g of strawberry jam) followed by a smoothie containing the powder. The Egg White Powder will be incorporated in the standardized smoothie containing water, fruits and chocolate/strawberry syrup totaling 250 Kcal. The total calories of the breakfast will be adapted to the calorie needs of each participant to account for 20-25% of their daily calorie intake.
  After a 9 h fast, blood will be taken before consumption of the standardized breakfast and smoothie (T= 0) and at 5, 10, 20, 30, 60, 90, 120, and 180 min after consumption of the smoothie. Participants will be given 15-25 minutes to eat their breakfast. Urine samples will be collected from participants before the smoothie consumption (0 h) and at 30 min, 90 min, 150 min, 6 hours, 12 hours, and 24 hours following consumption.

SUMMARY:
Bioactive peptides derived from food proteins show potential for improving human health. One of such promising peptides is namely IRW made from egg white hydrolysate and composed of three peptides. This is a feasibility study to assess the acute effect of IRW in egg white hydrolysate for the management of high sugar and blood pressure.

Participants at high risk of type 2 diabetes (T2D) or having T2D will undergo 4 consecutive treatments of 1 day each (randomly), during which they will consume a standardized breakfast with a smoothie containing different protein powders. Each treatment will be separated by a minimum of 1-week.

Participants in the healthy control group will undergo 1 treatment only (one day).

DETAILED DESCRIPTION:
Bioactive peptides derived from food proteins show vast potential for improving human health, in addition to providing nutritional value. One of such promising peptides is a short tripeptide IRW (made of three amino acids, isoleucine-arginine-tryptophan), the first discovered peptide that can activate ACE2 (angiotensin converting enzyme 2) preclinically. ACE2 is best known as the entry receptor of some coronaviruses, including the pandemic's SARS-CoV-2, while the primary role of ACE2 is to provide protection on the cardiometabolic system. Therefore, activation of ACE2 is a novel strategy to mitigate cardiometabolic diseases. A decade-long collaborative research on IRW has established a large body of knowledge about IRW's health effects on hypertension, type-2 diabetes (T2D)/insulin resistance (IR), oxidation, and inflammation. To translate the knowledge for human applications, it is essential to investigate the bioavailability and efficacy of bioactive peptide IRW in egg white hydrolysate.

IRW is derived from ovotransferrin, which accounts for ~12% of total egg white protein. Egg white powder without a process of hydrolyzation will not liberate the IRW, therefore, this will be used as a negative control. However, it is too costly to prepare IRW from pure ovotransferrin for functional food applications. To reduce the cost of production, whole egg white could be used as the starting material. IRW can only be released by a combination of thermolysin and pepsin. If only thermolysin is applied, a pentapeptide IRWCT is formed; as pepsin is naturally secreted in the stomach, egg white hydrolysate will be prepared using thermolysin. It is expected that IRW will be released in vivo by the gastrically secreted pepsin.

This study is the first to translate a peptide ACE2 activator as a functional food for human applications against metabolic syndrome (MetS, hypertension, T2D/Insulin Resistance). A functional food containing IRW provides a dietary strategy for the mitigation of metabolic syndrome and presents a value-added opportunity for the Canadian egg industry.

ELIGIBILITY:
Inclusion Criteria:

Healthy control group:

* Men and women aged between 18 and 70 years living in Edmonton (or Edmonton area/driving distance).
* Normal weight (BMI below 25 kg/m2 or Asian population below 23 kg/m2 )
* Waist circumference below the following ethnic specific cut offs: Canada / USA: <102 cm men and <88 cm women; Europids, Middle-Eastern, Sub-Saharan African, and Mediterranean: <94 cm men and <80 cm women; Asians, Japanese, South and Central Americans: <90 cm men and <80 cm women
* Fasting glucose <5.6 mmol/L
* HbA1c <5.6 %
* Blood pressure <130/85 mmHg
* Triglycerides <1.7 mmol/L
* HDL-Cholesterol >1.03 mmol/L men and >1.29 mmol/L women
* Body weight stable (within 3% fluctuation) for at least 6 months prior to the study
* Individuals who have never smoke, have smoke less than 100 cigarettes in their life or who are long term quitter (quit smoking a year or more ago)

Individuals at risk of diabetes/having type 2 diabetes:

* Men and women aged between 18 and 70 years living in Edmonton (or Edmonton area/driving distance).
* Overweight or obesity (BMI above 25 kg/m2 or Asian population above 23 kg/m2)
* Waist circumference at or above the following ethnic specific cut offs: Canada / USA: ≥ 102 cm men and ≥ 88 cm women; Europids, Middle-Eastern, Sub-Saharan African, and Mediterranean: ≥ 94 cm men and ≥ 80 cm women; Asians, Japanese, South and Central Americans: ≥ 90 cm men and ≥ 80 cm women
* Fasting glucose ≥ 6.0 mmol/L
* HbA1c ≥ 6.0 %
* Body weight stable (within 3% fluctuation) for at least 6 months prior to the study
* Individuals who have never smoke, have smoke less than 100 cigarettes in their life or who are long term quitter (quit smoking a year or more ago)

Exclusion Criteria:

* Individuals with a previous history of CVD, renal disorder, monogenic dyslipidemia, with endocrine disorders other than T2D
* Individuals taking chronic anti-inflammatory drugs (including aspirin, antihistamines, and omega-3 supplements)
* Pregnant/lactating women
* Individuals aged above 70 years
* Smokers (current smokers: daily/occasional and those who have smoked more than 100 cigarettes in their life)
* Individuals with specific nutritional restrictions (e.g. vegetarianism excluding eggs from their diet, vegan or with egg allergy) will be excluded
* Individuals with poorly controlled (HbA1c >12.0%) diabetes or taking exogenous insulin will be excluded. Other anti-diabetic and lipid-lowering medications will be documented.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2026-01-07 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Plasma Peptide concentration (IRW) overtime | 5, 10, 20, 30, 60, 90, 120, and 180 minutes after consumption of the smoothie
  iAUC for the plasma peptide concentration (IRW) after the test treatments compared to negative control smoothie

SECONDARY OUTCOMES:
Plasma glucose over time | 30, 60, 90, 120, and 180 minutes after consumption of the smoothie
  iAUC for plasma glucose (up to T= 180 minutes)
Plasma Insulin over time | 30, 60, 90, 120, and 180 minutes after consumption of the smoothie
  iAUC for plasma insulin (up to T=180 minutes)
Blood pressure over time | 60, 120, and 180 minutes after consumption of the smoothie
  Acute effect on blood pressure during the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jianping Wu, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada